CLINICAL TRIAL: NCT01775566
Title: A Phase I Clinical Trial to Compare the Pharmacokinetics and Safety of Eperisone HCl SR Tablet 75mg and Myonal Tablet 50mgafter Oral Administration in Healthy Male Subjects.
Brief Title: Clinical Trial to Compare the Pharmacokinetics and Safety of Eperisone HCl SR Tablet 75mg and Myonal Tablet 50mg
Status: Completed | Type: Observational
Sponsor: NVP Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: NVP-EPT-PK-01
Record Dates: First submitted 2013-01-17; First posted 2013-01-25 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Eperisone SR tablet 75mg, Myonal 50mg: Eperisone SR tablet 75mg Myonal 50mg

SUMMARY:
The purpose of this study is to Evaluate and Compare Safety and Pharmacokinetic of the Eperisone HCl SR and Myonal in healthy Korean male adults.

DETAILED DESCRIPTION:
Myonal: Eperisone Hydrochloride (muscle relaxant)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects age between 20 and 55 singed informed consent

Exclusion Criteria:

* Hypotension or hypertension has a history of allergy reaction of this drug or other drugs

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: acute low back pain
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Auclast, Cmax | Eperisone SR 0-24h, Myonal 0-24hr

SECONDARY OUTCOMES:
AUCinf, Tmax, t1/2, Css,min, Tss,max | Eperisone SR 0-24hr, Myonal 0-24hr

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Y Ran, M.D.Ph.D, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Gyeonggi SMB Growth Accelerating Center, Suwon, Gyeonggi-do, South Korea